CLINICAL TRIAL: NCT00638846
Title: Multi-Center Evaluation Of Two Silicone Hydrogel Toric Contact Lenses
Brief Title: Performance of Two Silicone Hydrogel Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0801; CTOR-501
Record Dates: First submitted 2008-03-10; First posted 2008-03-19 (Estimated); Results first posted 2010-07-19 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Vision Correction
Keywords: toric contact lenses; vision; comfort; toric fit characteristics; slit lamp findings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A toric (Experimental): senofilcon A, daily wear, toric contact lens worn for two weeks
  Interventions: Device: senofilcon A toric
- balafilcon A toric (Active Comparator): balafilcon A, daily wear, toric contact lens worn for two weeks
  Interventions: Device: balafilcon A toric

INTERVENTIONS:
Device: senofilcon A toric — silicone hydrogel toric lens, worn daily for 2 wks (2wks replacement)
  Other Names: ACUVUE OASYS
  Arms: senofilcon A toric
Device: balafilcon A toric — silicone hydrogel toric lens, worn daily for 2 wks (2wks replacement)
  Other Names: PureVision Toric
  Arms: balafilcon A toric

SUMMARY:
Evaluation of the clinical performance of two toric contact lenses in a 2-week, single masked (subject), daily wear, randomized, bilateral, parallel group study.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 45 years of age.
* Sign Written Informed Consent (See separate document).
* Be an existing successful daily wear toric soft contact lens.
* Require a visual correction in both eyes (monovision or uniocular fitting is NOT allowed).
* Does not require presbyopic correction (can read J1 @ normal reading distance).
* Have a sphere requirement in the range -1.00 and -5.00D (-5.25D refractive)
* Have refractive astigmatism between 0.75D and 2.50D in both eyes.
* Achieve visual acuity of 20/30 or better in each eye with spherical distance correction.
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  * No amblyopia.
  * No evidence of lid abnormality or infection.
  * No conjunctival abnormality or infection.
  * No clinically significant slit lamp findings (i.e. stromal edema, vascularisation, infiltrates or abnormal opacities).
  * No other active ocular disease.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Clinically significant (Grade 3 or 4) corneal stromal haze, corneal vascularisation, tarsal abnormalities, bulbar hyperemia, limbal hyperemia, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Corneal staining Grade 3 in more than one region.
* Has had refractive surgery. Has had eye injury/surgery within 8 weeks immediately prior to enrolment for this study.
* Abnormal lacrimal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* Polymethyl methacrylate (PMMA) or Rigid Gas Permeable (RGP) lens wear in the previous 8 weeks
* Extended lens wear in last 3 months.
* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Diabetic.
* Infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* Pregnancy, lactating or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial or in last 60 days.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme YOung, MPhil PhD, Study Director
Locations (19):
- United States (19):
  - Camp Eye Care Clinic, North Little Rock, Arkansas
  - James R. Dugue, O.D., Mission Viejo, California
  - Executive Park Eye Care, Colorado Springs, Colorado
  - Dr. Ted Brink and Associates, Jacksonville, Florida
  - Grene Vision Group, Neodesha, Kansas
  - Advanced Eyecare, PC, Raytown, Missouri
  - Dr. James Brobst, Florence, New Jersey
  - Fine Eye Care Associates, Rochester, New York
  - Warren Ophthalmology Associates, Warren, Ohio
  - Selden Eyecare LLC, Kittanning, Pennsylvania
  - Nittany Eye Associates, State College, Pennsylvania
  - Dr. David W. Ferris and Associates, Warwick, Rhode Island
  - Dr. Larry Menning, Chamberlain, South Dakota
  - Wishnow-Sugar Vision Group, Katy, Texas
  - Dr. William Bogus, Salt Lake City, Utah
  - Midlothian Optometric Center, Midlothian, Virginia
  - The Eye Specialists, Ltd., Virginia Beach, Virginia
  - The Eye & Contact Lens Clinic, Bremerton, Washington
  - Matus Eyecare, Franklin, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Senofilcon A Toric: senofilcon A toric contact lens. Analysis includes participants that completed the study.
- Balafilcon A Toric: balafilcon A toric contact lens. Analysis includes participants that completed the study.
Period: Overall Study
Arm/Group | Senofilcon A Toric | Balafilcon A Toric
Started | 137 | 139
Completed | 133 | 133
Not Completed | 4 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — lens issue | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Total
Number analyzed (Participants) | 137 | 139 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.81 (6.99) | 30.13 (7.69) | 29.97 (7.33)
Gender [Number; unit: participants] — Gender of 2 subjects assigned to balafilcon A is unknown.
  participants
    Female | 91 | 92 | 183
    Male | 46 | 45 | 91

OUTCOME MEASURES:

1. Primary Outcome: Lens Orientation
Description: Proportion of eyes with lens orientation within 5 degrees of optimal
Time Frame: 1 minute after insertion
Population: Analysis was performed on participants who completed the study per protocol. The data represents 274 eyes that wore senofilcon A lenses and 278 eyes that wore balafilcon A lenses.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: eyes
Arm/Group | Senofilcon A Toric | Balafilcon A Toric
Number analyzed (Participants) | 133 | 133
Number analyzed (eyes) | 266 | 266
proportion of eyes | 0.77 | 0.66
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Alternative hypothesis is senofilcon A toric is superior to balfilcon A toric by having less degrees of rotation; Test type: Superiority or Other; Generalized Linear Model; Odds Ratio (OR) = 1.739, 97.4% CI 2-sided [1.136 to 1.739] — Odds ratio was senofilcon A toric / balafilcon A toric

2. Primary Outcome: Lens Stability
Description: Lens stability is measured as the amount of rotation induced from blink after the lens has settled.
Time Frame: 10-15 minutes after insertion
Population: Analysis was performed on participants who completed the study per protocol.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: eyes
Arm/Group | Senofilcon A Toric | Balafilcon A Toric
Number analyzed (Participants) | 133 | 133
Number analyzed (eyes) | 266 | 266
proportion of eyes | 0.89 | 0.88
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Alternative hypothesis is that senofilcon A toric is superior to balafilcon A toric by having less degrees of instability; Test type: Superiority or Other; Generalized Linear Model; Odds Ratio (OR) = 1.138, 97.4% CI 2-sided [0.624 to 1.138] — Odds ratio was senofilcon A toric/balafilcon A toric

3. Secondary Outcome: Time to Fit Lens
Description: Time required for the optometrist to fit the lens.
Time Frame: after lens insertion
Population: Analysis was performed on participants who completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Senofilcon A Toric | Balafilcon A Toric
Number analyzed (Participants) | 133 | 133
minutes | 6.2789 (0.2045) | 7.4095 (0.1994)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Alternative hypothesis is that senofilcon A toric is superior to balafilcon A toric by having less time required to fit; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -1.1307, 97.5% CI 2-sided [-1.1307 to -0.5680], Standard Error of Mean 0.2856 — The mean difference is calculated as senofilcon A toric minus balafilcon At toric

4. Secondary Outcome: Subjective Lens Vision
Description: A weighted combined score calculated from individual vision-related questions asked on a 1-5 scale: 1 = most negative response to 5 = most positive response was used to derive vision outcomes. >0 = satisfactory vision, < 0 = unsatisfactory vision. Analysis is performed on combined 1 week and 2 week data.
Time Frame: measured at 1 and 2 weeks
Population: Analysis was performed on participants who completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Senofilcon A Toric | Balafilcon A Toric
Number analyzed (Participants) | 133 | 133
units on a scale | 0.1942 (0.09637) | -0.1738 (0.09716)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Alternative hypothesis is that senofilcon A is superior to balafilcon A; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.3680, 97.4% CI 2-sided [0.07001 to 0.3680], Standard Error of Mean 0.1331 — The mean difference is calculated as senofilcon A toric minus balafilcon A toric

5. Secondary Outcome: Overall Corneal Staining
Description: National Eye Institute 0-3 Scale: Grade 0 = Normal, Grade 1 = Mild, superficial stippling, Grade 2 = Moderate, punctuate staining including superficial abrasion of the cornea, Grade 3 = Severe, abrasion or corneal erosion, deep corneal abrasion or recurrent erosion.
Time Frame: After 2 weeks use
Population: Analysis was performed on participants who completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Senofilcon A Toric | Balafilcon A Toric
Number analyzed (Participants) | 133 | 133
units on a scale | 0.0919 (0.0178) | 0.1607 (0.0178)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Alternative hypothesis is that senofilcon A toric is superior to balafilcon A toric by having a lower grade fo corneal staining; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is -0.4; Mixed Models Analysis; Mean Difference (Final Values) = -0.0688, 97.5% CI 2-sided [-0.0688 to -0.0197], Standard Error of Mean 0.1648 — The mean difference is calculated as senofilcon A toric minus balafilcon A toric

6. Primary Outcome: Subjective Comfort
Description: Subjective comfort was derived from a weighted combined score calculated from individual comfort-related questions asked on a 1-5 scale: 1 = most negative response to 5 = most positive response. >0 = comfortable, < 0 = uncomfortable. Combined measures from Week 1 and Week 5.
Time Frame: 2 weeks of lens wear
Population: Analysis was performed on participants who completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Senofilcon A Toric | Balafilcon A Toric
Number analyzed (Participants) | 133 | 133
units on a scale | 0.1942 (0.09637) | -0.1738 (0.09716)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Alternative hypothesis is that senofilcon A toric is superior to balafilcon A toric; Test type: Superiority or Other; Mixed Models Analysis; Median Difference (Final Values) = 0.3680, 97.4% CI 2-sided [0.07001 to 0.3680], Standard Error of Mean 0.1331 — The mean difference is calculated as senofilcon A toric minus balafilcon A toric

ADVERSE EVENTS:
Arm/Group | Senofilcon A Toric | Balafilcon A Toric
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/133
Other Adverse Events (participants affected / at risk) | 0/133 | 0/133

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.